CLINICAL TRIAL: NCT01401140
Title: Coronary Surgery: Comparing the Protective Effects of Two Cardioplegic Solutions: Custodiol Versus St Thomas, on Cardiac Metabolism, as Assessed Using Microdialysis
Brief Title: Comparing the Protective Effects of Two Cardioplegic Solutions, on Cardiac Metabolism, as Assessed Using Microdialysis
Acronym: Cardioplégie
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Association AIRE (FR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0908033; 2009-A00506-51 (Other: Afssaps)
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Stenosis
Keywords: Coronary Artery Bypass; Coronary Artery Surgery; Coronary Artery Bypass Graft; Coronary Revascularization; Cardiac microdialysis; Custodiol; St Thomas; Cardioplegic solutions
MeSH Terms: conditions — Coronary Stenosis | interventions — St. Thomas' Hospital cardioplegic solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- St Thomas (Active Comparator)
  Interventions: Drug: St Thomas
- Custodiol (Experimental)
  Interventions: Drug: Custodiol

INTERVENTIONS:
Drug: St Thomas — Once the upper aorta has been clamped, the cardioplegic solution St Thomas will be administered directly into it via an anterograde approach. St Thomas will be infused every 30 minutes at a dosage of 10ml/kg bodyweight (infusion takes about three minutes). If the heart appears to be starting again (ventricular fibrillation) for more than three minutes, infusion will be resumed at the same rate until the heart is effectively stopped.
  Other Names: St Thomas solution or SLF 103 (Aguettant)
  Arms: St Thomas
Drug: Custodiol — Once the upper aorta has been clamped, the cardioplegic solution Custodiol will be administered directly into it via an anterograde approach. Custodiol will be injected in one bolus (20 ml/kg), which takes eight minutes. If the heart appears to be starting again (ventricular fibrillation) for more than three minutes, infusion will be resumed at the same rate until the heart is effectively stopped.
  Other Names: Custodiol (Eusa Pharma)
  Arms: Custodiol

SUMMARY:
An estimated 8% to 15% of patients hospitalized for a coronary pathology undergo coronary revascularization surgery with extracorporeal circulation (ECC). (1) Like most major cardiac surgical interventions, it is performed with the heart stopped; this leads to more or less severe myocardial ischemia. The heart is stopped (and therefore deprived of oxygen) for a duration that varies depending on the number of bypasses required, and on the local difficulties encountered. On average, myocardial ischemia lasts between 20 and 80 minutes. Heart protection during coronary revascularization surgery remains a crucial factor in limiting the heart's aerobic function during aortic clamping, and in minimizing the resulting post-operatory ventricular dysfunction. Its quality is a determining factor of the post-operatory issue.

High-performance heart protection solutions such as Custodiol have been used by heart surgeons for a few years. They are used as an alternative choice to other cardioplegic solutions, the efficacy of which has already been proven (St Thomas). These two myocardial protection solutions have never been evaluated in an in vivo, randomized, comparative trial.

DETAILED DESCRIPTION:
Myocardial microdialysis is the state-of-the-art technique for evaluating the protective effects of cardioplegic solutions; it enables physicians to monitor oxidation-reduction muscle metabolism during an ongoing operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient was referred to the Cardiovascular Surgery Unit for surgical coronary revascularization
* Patient has anterior interventricular stenosis
* Patient signed the informed consent form
* Patient is covered by health insurance

Exclusion Criteria:

* Patients with beating heart surgery indication (no extracorporeal circulation required)
* Emergency surgery and patients who suffered myocardial infarction less than a week before surgery
* Iterative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Lactate concentrations per-operatory | Every 10 minutes between the beginning of surgery, and declamping (per-operatory)
  Mean interstitial lactate concentrations (lactate peak and lactate/pyruvate ratio) observed between the beginning of surgery, and declamping in each patient group (St Thomas cardioplegia group vs Custodiol cardioplegia group)

SECONDARY OUTCOMES:
Anoxic variations 24h | Every hours after end of surgery and until the 24th hour following declamping.
  Interstitial lactate and pyruvate concentrations, lactate/pyruvate ratio, and glycerol concentration (glycerol is a marker of cell membrane damage),
Drug consumption | At 72 hours after declamping
  Inotropic drug consumption (dobutamin, noradrenalin, adrenalin) during the first 72 hours following declamping

CONTACTS AND LOCATIONS:
Overall Officials: Marco VOLA, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Eienne, Saint-Etienne, France